CLINICAL TRIAL: NCT05380557
Title: ARTEMIS: A Prospective Study of Patients With Early Stage Pancreatic Cancer Who Have Undergone Genetic Testing
Brief Title: ARTEMIS: Study of Patients With Early Stage Pancreatic Cancer Who Have Undergone Genetic Testing
Acronym: ARTEMIS
Status: Terminated | Type: Observational
Why Stopped: Low site engagement and accrual
Sponsor: Invitae Corporation (Industry)
Collaborators: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: CR-001-15
Record Dates: First submitted 2022-04-01; First posted 2022-05-19 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer; Resectable Pancreatic Cancer
Keywords: germline genetic testing; oncology; pancreatic cancer; resectable pancreatic cancer; early stage pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples including EDTA tubes for germline testing, streck tubes for other analyses, and archival tissue sample from a previous biopsy or resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Germline Pathogenic Variant in non-BRCA/PALB2 Gene: Patients will receive germline testing and provide streck tube blood samples and archival tissue sample at baseline. After germline testing results have been generated and released, patients and clinicians will be contacted for survey completion at months: 1, 4, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60 and survival collection every 6 months during years 3-10 post germline testing.
  Interventions: Diagnostic Test: Germline genetic testing
- Strong family history of pancreatic cancer but no identifiable germline pathogenic variant: Patients will receive germline testing and provide streck tube blood samples and archival tissue sample at baseline. After germline testing results have been generated and released, patients and clinicians will be contacted for survey completion at months: 1, 4, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60 and survival collection every 6 months during years 3-10 post germline testing.
  Interventions: Diagnostic Test: Germline genetic testing
- Negative germline testing and absence of strong family history: Patients will receive germline testing and provide streck tube blood samples and archival tissue sample at baseline. After germline testing results have been generated and released, patients and clinicians will be contacted for survey completion at months: 1, 4, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60 and survival collection every 6 months during years 3-10 post germline testing.
  Interventions: Diagnostic Test: Germline genetic testing
- Pathogenic Variant in BRCA1/2 or PALB2: Patients will be offered enrollment into the sister trial, APOLLO (NCT04858334). Patients and clinicians will be contacted for survey completion at months: 1, 4, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60 and survival collection every 6 months during years 3-5.
  Interventions: Diagnostic Test: Germline genetic testing

INTERVENTIONS:
Diagnostic Test: Germline genetic testing — Germline genetic testing will be provided to each patient

SUMMARY:
This study includes participants with pancreatic cancer who are undergoing genetic testing at Invitae related to their diagnosis of pancreatic cancer.

Our goal in this study is two-fold. First, we would like to research whether any inherited changes in genes may be associated with pancreatic cancer. Second, we would like to learn more about patient experiences with genetic testing, such as patient understanding of the testing, health-related actions taken (or planned to take) as a result of testing, communication and action of family members based on test results, and psychological impact of testing.

This research study involves allowing collection of tumor tissue (from a prior biopsy and/or surgery), a blood sample, and sending surveys to participants for their opinion on the impact of the genetic testing as well as clinicians for relevant baseline and medical history information.

DETAILED DESCRIPTION:
Patients will be contacted for patient outcomes survey completion at months: 1, 4, 8, 12, 18, 24, 30, 36, 42, 48, 54, and 60. Patients will also be contacted for survival collection every 6 months during years 3-5 post germline testing.

Clinicians will be contacted for relevant medical history, treatment, and survival data at the same time points.

At baseline, 3 samples types will be collected: 1. EDTA tube for germline genetic testing. 2. Streck tubes for whole genome sequencing and other analyses. 3. Tumor block from surgical resection. If block is unavailable 10 unstained slides are an acceptable substitute.

ELIGIBILITY:
Inclusion Criteria:

* Patient has consented to germline genetic testing
* Patient has a histologically confirmed diagnosis of pancreatic cancer
* Patient has undergone or is planned to undergo surgical resection with curative intent
* Patient is willing to allow collection of a tissue sample from surgical resection
* Patient is willing to provide research blood samples (every 6 months for 2 years)
* Patient must be at least 18 years of age

Exclusion Criteria:

* Patient has evidence of metastatic or recurrent pancreatic cancer at time of consent
* Patient is unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with resectable pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Germline pathogenic variants identified on Invitae's 84 gene Multi Cancer panel | Will be assessed at baseline only.
Overall survival | Will be assessed in patient and clinician surveys distributed every 4 months for the first year post germline testing
Overall survival | Will be assessed every 6 months for years 2 - 10 post germline testing

CONTACTS AND LOCATIONS:
Locations (1):
- Invitae SF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Invitae may share de-identified information and data generated through the study with third parties, including biopharmaceutical companies and biomedical researchers (e.g. academic), for clinical trials, drug development, and other disease-related research purposes.
  Only a subset of Invitae personnel will have access to PHI. The PHI will be stored in a secure location and will only be made available to Invitae personnel involved in the Study. Any academic publication of data analysis from this Study will use de-identified information only.